CLINICAL TRIAL: NCT00667147
Title: Phase I Trial of Abraxane Administered on a Weekly and Three Weekly Schedule in Combination With Vandetanib
Brief Title: Phase I Abraxane Weekly and Three Weekly Schedule With Vandetanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: AstraZeneca (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0C-07-3
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Weekly Abraxane and Daily Vandetanib
- B (Experimental)
  Interventions: Drug: Abraxane every three weeks and daily vandetanib

INTERVENTIONS:
Drug: Weekly Abraxane and Daily Vandetanib — Abraxane once a week for three weeks, followed by one week with no Abraxane. Vandetanib once a day every day for 28 days. This four week period is called a cycle.
  Arms: A
Drug: Abraxane every three weeks and daily vandetanib — Abraxane on day one of study therapy, followed by 20 days of no Abraxane. Vandetanib once a day every day for 21 days. This three week period is called a cycle.
  Arms: B

SUMMARY:
This study uses the drugs Abraxane (also called ABI-007) and Vandetanib (also called Zactima and ZD6474). Abraxane has been approved by the Food and Drug Administration (FDA), for the treatment of breast cancer. Vandetanib is an experimental drug and has not been approved by the FDA for the treatment of any condition. Vandetanib has shrunk some non-small cell lung cancer, prostate cancer and thyroid cancer in some studies in humans. This combination of drugs is not approved for the treatment of any condition by the FDA.

This study is being done in two phases. The first phase of the trial has two main objectives: 1) To find the highest daily dose of vandetanib that can be given safely with once weekly Abraxane and 2) To find the highest daily dose of vandetanib that can be given safely with Abraxane given every three weeks. Participants will be randomly assigned (like flipping a coin) to receive Abraxane weekly (Arm A) or once every three weeks (Arm B). The dose of Abraxane given will remain the same for the whole study - 100 mg/m2 when given weekly and 260 mg/m2 when given every three weeks. Participants will be entered onto each arm of the study in groups of three, and higher doses of vandetanib will be given each group of participants. The increase of vandetanib will stop once more than one participant has serious side effects. The highest dose of vandetanib that can be given with Abraxane (without serious side effects) in each Arm will be called the pilot dose.

In the second phase of the study twenty participants will be randomly assigned to Arm A or Arm B and receive the pilot dose of vandetanib that was reached in the first phase of the study. The purpose of the second phase of the study is to see how many tumors shrink when participants receive the pilot dose of the drug combination on each Arm, as well as to gather more information about the side effects.

ELIGIBILITY:
Inclusion Criteria:

* SWOG performance status of 0-2
* Projected life expectancy of at least 3 months
* Female and or male age 18 years and over
* Provision of informed consent prior to any study-related procedures.
* Patients must not have history of torsades de pointes ventricular arrythmia
* Patients must not have a prolonged QT interval > 450 msec on baseline EKG in the presence of normal serum and magnesium values. Patients with QTc with Bazett's correction that is unmeasurable are ineligible. (Note: If a subject has a QTc interval less than or equal to 450 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <450 msec in order for the subject to be eligible for the study.) Patients who are receiving a drug that has a risk of QTc prolongation are excluded if QTc is ≥ 460 msec.
* Female patients must not be pregnant due to the potential mutagenicity and teratogenicity of this treatment. A pregnancy test must be administered 7 days prior to administration of therapy to women of childbearing potential.
* Patients must agree to use some form of contraception while on this study at initiation and for the duration of participation in the study. Sexually active males must also use a reliable and appropriate method of contraception. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Patients must have recovered from acute toxicities from previous surgery, chemotherapy or radiation therapy
* Adequate organ function defined as:

ANC > 1500/mm3 Platelet count > 100,000 cells/mm3 Hemoglobin > 9.0g/dL Serum creatinine < 1.5 mg/dl or creatinine clearance > 50 mL/minute Hepatic function: Patients must have adequate liver functions: AST or ALT < 2.5 X upper limit of normal (ULN), alkaline phosphatase < 2.5 X upper limit of normal. In patients with bone metastasis and no evidence of liver metastasis and bilirubin < upper limit of normal an alkaline phosphatase < 5 ULN will be allowed.

In patients with known liver involvement: AST or ALT and alkaline phosphatase < 5 ULN, Serum Bilirubin < 1.5 mg/dL

* Peripheral neuropathy grade 0-1
* No other concomitant therapy directed at the cancer is allowed. All prior therapy must have been completed > 4 weeks prior to study enrollment.
* Patients diagnosed with advanced prostate cancer must have progressed on or have been intolerant of a docetaxel based regimen.

Exclusion Criteria:

* Laboratory results:

  * Serum bilirubin > 1.5 the upper limit of reference range (ULRR)
  * Serum creatinine >1.5 x ULRR or creatinine clearance < 50 mL/minute (calculated by Cockcroft-Gault formula.)
  * Potassium, < 4.0 mmol/L despite supplementation; serum calcium (ionized or adjusted for albumin,) or magnesium out of normal range despite supplementation
  * Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
  * Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease >2 (see Appendix B) within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
  * History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
  * QTc prolongation with other medications that required discontinuation of that medication.
  * Congenital long QT syndrome,or 1st degree relative with unexplained sudden death under 40 years of age.
  * Presence of left bundle branch block (LBBB.)
  * Any concurrent medication that may cause QTc prolongation or induce Torsades de Pointes ( Protocol Appendix A lists relevant medications that have a risk of Torsades de Pointes or QTc prolongation.) Drugs listed in Appendix A, Table 2, that in the investigator's opinion cannot be discontinued, are allowed however, must be monitored closely (please see section 4.2).
  * Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
  * Currently active diarrhea that may affect the ability of the patient to absorb the Vandetanib or tolerate diarrhea.
  * Women who are currently pregnant or breast feeding.
  * Receipt of any investigational agents within 30 days prior to commencing study treatment
  * Last dose of prior chemotherapy discontinued less than 4 weeks before the start of study therapy
  * Last radiation therapy within the last 4 weeks before the start of study therapy, except palliative radiotherapy
  * Any unresolved toxicity greater than CTC grade 1 from previous anti-cancer therapy
  * Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy.
  * Previous enrollment in the current study.
  * Patients with the following conditions: Colon cancer, Rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-03; Primary Completion 2012-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | First Cycle of Study Therapy

SECONDARY OUTCOMES:
RECIST Response | Until Patient goes off study
Toxicity | Until Patient Goes off study

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, M.D., Principal Investigator — U.S.C. / Norris Comprehensive Cancer Center
Locations (1):
- University of Southern California (U.S.C.)/ Norris Comprehensive Cancer Center, Los Angeles, California, United States